CLINICAL TRIAL: NCT02659618
Title: Identification of Serum Biomarkers for CD15+ Hypodense Neutrophils in Severe Asthma
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mary Tobin, Director, Rush University Medical Center
Other Study IDs: ML29345
Record Dates: First submitted 2015-07-06; First posted 2016-01-20 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2020-12

CONDITIONS: Severe Persistent Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood and serum will be drawn and shipped to Genentech for analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe Persistent Asthma: All subjects will have severe persistent asthma diagnosed by a doctor.

SUMMARY:
The goal of this study is to identify a serum biomarker(s) that can detect increased levels of a population of CD15+ hypodense neutrophils termed low-density granulocytes (LDG) in the blood of patients with severe persistent asthma.

DETAILED DESCRIPTION:
Neutrophils are implicated in the pathophysiology of multiple asthma phenotypes. It was shown in study IST Q4935s that low-density granulocytes (LDG) are elevated in the blood of patients with moderate or severe asthma. The greatest frequency and the highest percentages of LDG were observed in subjects with severe asthma. The LDG, which were first identified and characterized in systemic lupus erythematosus (SLE) patients, have been reported to display increased cytotoxicity for endothelial cells, increased tendency to form neutrophil extracellular traps, and increased production of tumor necrosis factor (TNF). It was also observed that the LDG expressed increased levels of CD15, which can facilitate attachment of activated platelets to the LDG. Identification of a putative serum biomarker that correlates with increased levels of the CD15+ LDG may be useful for the detection of neutrophil-associated inflammation in severe asthma.

Thirty subjects will be screened to identify 20 subjects with severe persistent asthma. The following data and/or samples will then be obtained within three weeks of the clinical assessment: (1) the percentages of LDG will be quantified by flow cytometry; (2) a blood sample will be collected into a PAXgene Blood tube and stored until shipped to Genentech for gene profiling analysis; and (3) a serum sample will be collected for measurement of total immunoglobulin E (IgE) and for future confirmation of potential biomarkers identified in the gene profiling analyses.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of severe persistent asthma;
* Positive skin test or radioallergosorbent test (RAST) for an aeroallergen;
* Male or female age 12-65 years;
* Non-smoker.

Exclusion Criteria:

* Asthma exacerbation requiring treatment with or increase in oral corticosteroids within 30 days prior to the study;
* Respiratory infection within 30 days prior to the study;
* Starting or requiring a change in allergen immunotherapy within 30 days prior to the study;
* Having been treated with Xolair within the past year;
* Requiring chronic immunosuppressive therapy;
* Having taken methotrexate, gold salts, cyclosporine, or macrolide antibiotics within 3 months prior to study;
* Having taken an investigational drug within 30 days prior to the study;
* Have a history of drug or alcohol abuse;
* Pregnancy

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thirty prospective subjects will be screened to identify 20 subjects with severe persistent asthma. These subjects will be recruited from the Allergy/Immunology outpatient clinic at Rush University Medical Center along with self-referral through advertising posted on campus.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Percentage of low density granulocytes (LDG) in the peripheral blood mononuclear cell (PBMC) | Visit 1 day
mRNA levels in severe asthmatics as analyzed by gene profiling analysis | Visit 1 day
  Messenger ribonucleic acid (mRNA) expression levels for blood leukocyte proteins.

SECONDARY OUTCOMES:
Number of Participants with elevated LDG levels in severe asthmatics using gene profiling analysis on a single PAXgene tube sample | Visit 1 day
Serum samples will be collected and analyzed for measurement of total IgE | Visit 1 day
  Correlation between LDG in severe asthma and biomarkers identified in gene profiling analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University Consultants in Allergy/Immunology, Chicago, Illinois, United States